CLINICAL TRIAL: NCT06198231
Title: Effects of Pilates Exercises on Balance and Gait in School Going Children
Brief Title: Effects of Pilates Exercises on Balance and Gait in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0758
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Children
Keywords: Balance; Pilates exercises; Postural control; Randomized control
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises (Experimental): The experimental group will receive the same program of exercises given to the control group, 45 minutes of Pilates exercises (such as back twists, single leg circles, standing splits, alternate toe touches, ball leg lifts).The Pilates exercises will be aimed at improving lower-limb strength, flexibility, and coordination, and they will be performed on a mat, using a medical ball. The focus will be on maintaining core contraction, spinal and pelvic alignment, and respiration rhythm. Ten repetitions of Pilates exercises will be performed, with a 2-minute rest period between repetitions.
  Interventions: Other: Pilates exercises
- Flexibility ,strength and endurance excercises (Active Comparator): Control group will perform flexibility exercises for the hip (flexors and adductors), knee (flexors and extensors), and calf muscle, with a hold of 15 sec ,5 repetitions. Strengthening exercises for core muscles (curl-ups, prone extension),hip extensors (in prone position), hamstrings, quadriceps (knee extension in high sitting).Walking in all directions, standing on rough and soft surfaces, stepping down and up, walking,standing on one limb with both eyes closed and open. Each session will start with a 5-minute warm-up and 5-minute cool-down, session duration 45 minutes,3 times a week.
  Interventions: Other: Flexibility ,strength and endurance excercises

INTERVENTIONS:
Other: Pilates exercises — Pilates exercises
  Arms: Pilates exercises
Other: Flexibility ,strength and endurance excercises — flexibility ,strength and endurance excercises
  Arms: Flexibility ,strength and endurance excercises

SUMMARY:
The school children often spend prolonged hours in sedentary activities and may not engage in sufficient physical exercise A sedentary lifestyle among school-going children is a growing concern in modern society. Children are spending more time sitting down and less time being physically active. This can lead to a variety of health problems, including obesity, poor posture, and a lack of cardiovascular fitness. Postural control is crucial for children's balance, gait, and functional tasks, and core stability and hip muscle strength play significant roles in maintaining proper posture and facilitating movement. Pilates is a popular exercise program known for improving core strength, balance, flexibility, and posture. Understanding the potential benefits of Pilates exercises on muscle strength and postural control in this population is essential, considering the sedentary lifestyles of many school children. Limited research has examined the effectiveness of Pilates exercises in school-aged children This randomized controlled trial will be conducted in schools in Daska City Govt. girls high school Raj okay Tehsil DASKA, Govt Girls elementary school KOT JANDHU Tehsil DASK e.g over a duration of six months. The sample size will consist of 96 children aged 6 to 9 years, divided equally into a control group and an experimental group. The inclusion criteria specify children without acute illnesses or injuries, within the normal BMI range, and free from cognitive impairments or chronic medication use. The control group will receive exercises that will focus on flexibility, strength, and endurance targeting postural stability for 45 minutes, while the experimental group will receive program of exercises including 15 minutes of conventional exercise along(strengthening, flexibility exercises) with 30 minutes of Pilates excercises including ( back twists, single leg circles, standing splits, alternate toe touches, ball leg lifts) for 3 times a week, of Pilates exercises aimed at improving lower-limb strength, flexibility, and coordination. Assessments will be conducted at baseline, 4th week, and 8th-week using measures such as the Pediatric Berg Balance Scale, walking speed assessment, FRT.

DETAILED DESCRIPTION:
The sample size will consist of 96 children aged 6 to 9 years, divided equally into a control group and an experimental group. The inclusion criteria specify children without acute illnesses or injuries, within the normal BMI range, and free from cognitive impairments or chronic medication use. The control group will receive exercises that will focus on flexibility, strength, and endurance targeting postural stability for 45 minutes, while the experimental group will receive program of exercises including 15 minutes of conventional exercise (strengthening, flexibility exercises) along with 30 minutes of Pilates exercises including ( back twists, single leg circles, standing splits, alternate toe touches, ball leg lifts) for 3 times a week. Each session will be started with a 5-minute warm-up and concluded with a 5-minute cool-down. Pilates exercises aimed at improving lower-limb strength, flexibility, and coordination. Assessments will be conducted at baseline, 4th week, and 8th-week using measures such as the Paediatric Berg Balance Scale, walking speed assessment, FRT. This randomized controlled trial will be conducted in schools in Daska City Govt. girls high school Raj okay Tehsil DASKA, Govt Girls elementary school KOT JANDHU Tehsil DASK e.g over a duration of six months.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 and 9 years
* Both male and female students.
* Students with normal BMI.
* Students willingness for participation.

Exclusion Criteria:

* Students with cognitive impairments.
* Students with conditions such as chronic fatigue, myalgia, limb deformity or any orthopedic condition.
* Students who are currently taking any form of medication for chronic illnesses.
* Students with limb deformities e.g flat foot, genuvelgum, genuvarum and leg length discrepancy.
* Students with any type of psychological problem.
* Children who have participated in similar Pilates or physical therapy exercise programs targeting balance and gait in the past six months

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
pediatric berg balance scale | 8 weeks
  The Pediatric Balance Scale (PBS) is an assessment tool consists of 14 different balance tasks that challenge various aspects of balance control, including static and dynamic balance (6) The tasks involve different postural positions, such as sitting, standing, and transferring weight, and may require the child to maintain balance while performing specific movements or tasks. Intra class correlation coefficient (ICC) = 0.998] or individual items (Kappa Coefficients, k = 0.87 to 1.0)
walking speed assessment | 8 weeks
  The walking speed assessment will utilize a 6-minute walk test in which the child will be instructed to walk back and forth in a designated hallway for 6 minutes. They will pivot briskly around cones without hesitations. Participants will be accompanied by the assessor, who will be positioned just behind them without leading or influencing their walking speed. The assessment will be conducted before and after the exercise intervention to assess improvements in basic mobility. Strong test-retest reliability was demonstrated (intra class correlation = 0.97).

SECONDARY OUTCOMES:
functional reach test | 8 weeks
  The test involves the participant standing next to a wall, with their arm at 90 degrees of shoulder flexion and a closed fist. The starting position is recorded, and the participant is instructed to reach forward as far as possible without taking a step. The distance between the starting and ending positions is measured and recorded. Three trials will be performed, and the average of the last two trials will be noted. The reach distance is typically measured in inches. The criteria for stopping the test include the patient's feet lifting off the floor or falling forward. The intra-class correlation coefficient range 0.90 - 0.97).

CONTACTS AND LOCATIONS:
Overall Officials: kirn arshad, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franco MR, Grande GHD, Padulla SAT. Effect of pilates exercise for improving balance in older adults (PEDro synthesis). Br J Sports Med. 2018 Feb;52(3):199-200. doi: 10.1136/bjsports-2016-097073. Epub 2016 Nov 4. No abstract available. PMID 27815239